CLINICAL TRIAL: NCT03092570
Title: Assessment of Cerebellar Stimulation Effect on Motor Learning in Ageing Population and Stroke Patients
Brief Title: Manual Dexterity Control After Cerebellar Stimulation
Acronym: MADECCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D16-P03
Record Dates: First submitted 2017-02-15; First posted 2017-03-28 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Stroke
Keywords: Motor learning; stroke; tDCS; upper limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- tDCS Post-CVA (Experimental): The participants will get a 20min stimulation at a maximal intensity of 2mA
  Interventions: Device: With stimulation
- Sham Post-CVA (Sham Comparator): The tDCS will be placed as for the Experimental group and will last 30 seconds at the beginning of task
  Interventions: Device: No stimulation
- tDCS Young Healthy (Experimental): The participants will get a 20min stimulation at a maximal intensity of 2mA
  Interventions: Device: With stimulation
- Sham Young Healthy (Sham Comparator): The tDCS will be placed as for the Experimental group and will last 30 seconds at the beginning of task
  Interventions: Device: No stimulation
- tDCS Older Healthy (Experimental): The participants will get a 20min stimulation at a maximal intensity of 2mA
  Interventions: Device: With stimulation
- Sham Older Healthy (Sham Comparator): The tDCS will be placed as for the Experimental group and will last 30 seconds at the beginning of task
  Interventions: Device: No stimulation

INTERVENTIONS:
Device: With stimulation — ramp stimulation from 0 to 2 mA followed by 20 minutes of stimulation at 2mA while practicing during 3 of the 4 sessions
  Arms: tDCS Older Healthy; tDCS Post-CVA; tDCS Young Healthy
Device: No stimulation — ramp stimulation from 0 to 2 mA followed by 30 sec of stimulation at 2mA.
  Arms: Sham Older Healthy; Sham Post-CVA; Sham Young Healthy

SUMMARY:
This study will assess the putative advantages of cerebellar stimulation on motor learning abilities of stroke patients. In order to have a control group to refer to, the effect of cerebellar stimulation on healthy young and old participants will also be assessed.

DETAILED DESCRIPTION:
Cerebrovascular accidents (CVA) are the first cause of acquired disability in France. Despite rehabilitation interventions, a great proportion of patients suffers from motor disability in the upper limb. Recently, several studies have shown that post CVA patients exhibit great neural plasticity as a direct consequence of their condition.

Interestingly, the transcranial direct current stimulation (tDCS) is a non-invasive electro stimulation technique that allows for a modulation of cerebral activity. It has been shown that when applied to the cerebellum, tDCS increases learning performances of healthy subjects. Yet, motor rehabilitation after a CVA highly relies on motor (re)learning. The cerebellar tDCS thus appear as a promising method to enhance the performance of post-CVA motor learning and consequently the benefits of post-CVA rehabilitation.

The current study aims to promote the post CVA neural plasticity by using the tDCS in order to enhance motor learning of the upper limb.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Affiliated to the French health insurance or similar organisation
* Signed informed consent
* Clinical examination

For "Post-AVC patients" :

* at least 18 years old
* completed the Moberg Pick-up test with a minimum score of 20 secondes For "Young healthy" group
* 18 = or > years = or <30 For "Older healthy" group
* 50 > or = years = or < 80

Exclusion Criteria:

* Metallic implant in the head
* Pacemaker, or other electronic implanted devices
* Other central neurological disease
* Pregnancy, breast feeding
* Previous history of neurosurgery or seizures or 1st degree relative with history of seizures
* History of medical neurological or psychiatric disorders
* Participation to another study using cerebral stimulation
* History of bi-polar or recurring depressive disorders
* Planned carotid revascularization, severe caridac disease
* Kidney failure (transaminase > 2 times normal value)
* Other invalidating condition or deficiency interfering with the study

For "Post-AVC patients" :

* NIHSS score > 20
* Cerebellar ischemic CVA

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Force control | Day 1
  Measurement in Newton of the force applied by each finger.
Force control | Day 2
  Measurement in Newton of the force applied by each finger.
Force control | Day 3
  Measurement in Newton of the force applied by each finger.
Force control | Day 10
  Measurement in Newton of the force applied by each finger.
Overflow | Day 1
  Measurement in ms of the involuntary finger movements.
Overflow | Day 2
  Measurement in ms of the involuntary finger movements.
Overflow | Day 3
  Measurement in ms of the involuntary finger movements.
Overflow | Day 10
  Measurement in ms of the involuntary finger movements.

SECONDARY OUTCOMES:
Moberg Pick-up Test | Day 1
  Assessment of the functionality of the hand. One score will be given at the end of the test.
Moberg Pick-up Test | Day 2
  Assessment of the functionality of the hand. One score will be given at the end of the test.
Moberg Pick-up Test | Day 3
  Assessment of the functionality of the hand. One score will be given at the end of the test.
Moberg Pick-up Test | Day 10
  Assessment of the functionality of the hand. One score will be given at the end of the test.
Action Research Arm Test | Day 1
  Assessment of the upper limb mobility. One score will be given at the end of the test
Action Research Arm Test | Day 2
  Assessment of the upper limb mobility. One score will be given at the end of the test
Action Research Arm Test | Day 3
  Assessment of the upper limb mobility. One score will be given at the end of the test
Action Research Arm Test | Day 10
  Assessment of the upper limb mobility. One score will be given at the end of the test
Finger time release | Day 1
  Time needed to release the finger force when needed (in ms).
Finger time release | Day 2
  Time needed to release the finger force when needed (in ms).
Finger time release | Day 3
  Time needed to release the finger force when needed (in ms).
Finger time release | Day 10
  Time needed to release the finger force when needed (in ms).

CONTACTS AND LOCATIONS:
Overall Officials: Florence COLLE, MD, Principal Investigator — CHSA
Locations (2):
- France (2):
  - Centre de Recherche Clinique (CRC) - CHSA, Paris
  - Service de Médecine Physique et Rédaptation, Paris

IPD SHARING:
Plan to Share IPD: No